CLINICAL TRIAL: NCT01410292
Title: Glycemic and Satiety Response to Meals With Different Fiber Content and Glycemic Index in Type 2 Diabetic Patients
Brief Title: Glycemic and Satiety Response to Fiber and Glycemic Index of Meals in Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Mirela Jobim de Azevedo, Endocrine Division of Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: GPPG 10-0472
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: fiber; glycemic index; glycemic response; diabetes; ghrelin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Meals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- meal D (Experimental): low fiber and low GI
  Interventions: Other: GI and fiber meals; Other: meals
- meal C (Experimental): low Fiber and High GI
  Interventions: Other: GI and fiber meals; Other: meals
- meal B (Experimental): high Fiber and low GI
  Interventions: Other: GI and fiber meals; Other: meals
- meal A (Experimental): high fiber and high GI meal
  Interventions: Other: GI and fiber meals; Other: meals

INTERVENTIONS:
Other: GI and fiber meals — meals with different fiber content and glycemic index
Other: meals — four different meal regarding GI and fiber content

SUMMARY:
The aim of this study is to assess the post-prandial response of four breakfast with different content of dietary fiber and glycemic index on glycemic response and satiety in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Design study:

Single-blind crossover randomized clinical trial

Hypothesis:

A meal with high GI and high fiber content determines a lower glycemic response compared to a meal with high GI and low fiber content (fiber beneficial effect on glycemic response independent of glycemic index.

Test meals:

Four test meals isocaloric and with the same proportion of macronutrients will be evaluated (5 kcal/kg, 17% of energy provided by protein, 58% of energy provided by carbohydrates, and 25% of energy provided by fat):

Test Meal A:high glycemic index (GI= 60.3%) and high fiber content(5.88g) Test Meal B:high glycemic index (GI= 62.8%) and LOW fiber content(2.05g) Test Meal C:low glycemic index (GI= 37.0%) and high fiber content(5.75g) Test Meal D:low glycemic index (GI= 38.4%) and high fiber content(1.91g)

Outcomes:

Glycemic response: serum glucose and insulin Satiety response: serum ghrelin and subjective assessment of satiety by a specific scale for measurement of appetite in single test meal studies.

Logistic:

Patients will undergo a clinical, nutritional and laboratory evaluation for confirm the inclusion criteria and will be request to give their written informed consent.

All participants will test each meal with a mean of seven days separating the individual test days.A 12h fast will precede all the study visits.Pre-and postprandial blood samples will be draw to determine the concentrations of serum insulin and plasma glucose, and ghrelin through an antecubital cannula before and 15, 30, 45, 60, 90, 120 and 180 min after the test meals. The VAS scale will be applied in these times.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes,
* HbA1c < 9%,
* BMI < 35kg/m²,
* Metformin and/or diet as treatment for diabetes

Exclusion Criteria:

* Use of insulin as diabetes treatment
* digestive disease with malabsorption
* diabetes neuropathy with gastroparesis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-09 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
glycemic control | fasting and post-prandial (differents times during 180 minutes)
  glucose and insulin

SECONDARY OUTCOMES:
measures of satiety and appetite | fasting and post-prandial (different times for 180 min)
  ghrelin and subjective analogue scale of appetite

CONTACTS AND LOCATIONS:
Overall Officials: Flávia M Silva, Study Chair — Hospital de Clínicas de Porto Alegre; Thais Steemburgo, Study Chair — Hospital de Clínicas de Porto Alegre; Caroline Kramer, Study Chair — Hospital de Clínicas de Porto Alegre; Giovana Menegotto, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Silva FM, Kramer CK, Crispim D, Azevedo MJ. A high-glycemic index, low-fiber breakfast affects the postprandial plasma glucose, insulin, and ghrelin responses of patients with type 2 diabetes in a randomized clinical trial. J Nutr. 2015 Apr;145(4):736-41. doi: 10.3945/jn.114.195339. Epub 2015 Feb 11. PMID 25833777